CLINICAL TRIAL: NCT05323773
Title: How is Calf Muscle Endurance Related to Ankle Injuries in TeamGym Athletes?
Status: Completed | Type: Observational
Sponsor: Susanne Beischer (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Susanne Beischer, Principal Investigator, Göteborg University
Organization: Göteborg University (Other)
Other Study IDs: Projektfot1
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ankle Injuries; Foot Injury; Overuse Injury; Ankle Sprains
Keywords: Gymnastics; TeamGym; Muscular Fatigue; Muscular Endurance
MeSH Terms: conditions — Ankle Injuries; Foot Injuries; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specific aims of this study are to:

* describe how many heel raises and side hops TG athletes of various ages can perform and how far they can jump, one leg at a time.
* examine how calf muscle endurance and hop performance are related to the risk of new injuries in the foot, ankle, and lower leg in TG athletes.

The investigators hypothesise that atletes with superior performance in the tests for muscular endurance and hop performance will report fewer injuries during the follow up period.

DETAILED DESCRIPTION:
TeamGym (TG) is the most common gymnastics discipline in Sweden. There is a relatively high injury incidence of 2,2-3,4 injuries per 1000 hours of gymnastic activity. Muscular fatigue has been proposed as a risk factor for sustaining an injury in gymnastics, but this has yet not been examined.

In TG, the lower extremity is more susceptible to injuries than the spine and upper extremity, with injury rates ranging between 60 - 77% for the lower extremity. More specifically, the foot, ankle, and the lower leg account for 40 - 56% of all reported injuries, consisting mostly of ankle injuries.

In clinical and research settings, heel raises and side hops are commonly used to assess muscular endurance in the lower leg. Furthermore, it is common to also include a hop performance test to assess the physical capacity of an athlete following an injury to the foot, ankle, or lower leg. However, there are normative values published of the aforementioned tests, in TG athletes

The overall purpose of this project is to facilitate and improve the caretaking of TG athletes who have sustained various types of injuries in the foot, ankle and lower leg.

Specific aims are to:

* describe how many heel raises and side hops TG athletes of various ages can perform and how far they can jump, one leg at a time.
* examine how calf muscle endurance and hop performance are related to the risk of new injuries in the foot, ankle, and lower leg in TG athletes.

The investigatorshypothesise that atletes with superior performance in the tests for muscular endurance and hop performance will report fewer injuries during the follow up period.

About 200 athletes who regulary participate in TeamGym training (at least once per week) and understand written and spoken Swedish will be included in this study.

Athletes with a recent injury to the foot, ankle, or lower leg or the presence of with other injuries to the lower limb or spine that may be accentuated or affect test results will be excluded.

Data regarding numbers of new injuries (acute and overuse injuries) in the foot, ankle and/or lower leg within six months after baseline testing aswell as severity score of the overuse injuries will be measured bi-weekly with the Oslo Sports Trauma Research Center (OSTRC) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Regular participation in TeamGym training (at least once per week)
* Understanding written and spoken Swedish

Exclusion Criteria:

* Recent (defined as: in the last 4 weeks before baseline testing) injury to the foot, ankle, or lower leg = exclusion from hop tests.
* Presence of other injuries to the lower limb or spine that may be accentuated or affect test results.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: TeamGym athletes (members of the Swedish Gymnastics Federation) in Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
New injury | Within six months after baseline testing.
  Number of new acute/overuse injuries in the foot, ankle or lower leg.

SECONDARY OUTCOMES:
Severity of overuse injury | Bi-weekly follow-ups over a 6 month period.
  Answers from 4 questions regarding severity are scored from 0 to 25, and summed to calculate a severity score between 0 (= no problems) and 100 (= maximum level of problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
One of the purposes of the project is describing normative data regarding muscular endurance and hop performance in TeamGym athletes and the results will therefore be published. Thus, there will be no need to make IPD available for other researchers.